CLINICAL TRIAL: NCT01028859
Title: Phase I Clinical Trial to Assess the Safety and Pharmacokinetic Profile of CKD-516 in Patients With Advanced Solid Cancers Failed to Standard Therapy
Brief Title: Safety Study of Increasing Doses of CKD-516 in Patients With Advanced Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Chong Kun Dang Pharmaceutical, Medical Department
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 127ASC09E
Record Dates: First submitted 2009-12-03; First posted 2009-12-09 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2009-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Tubulin polymerization inhibitor; CKD-516; Phase I; Vascular disrupting agent; DCE MRI
MeSH Terms: interventions — N-(4-(3-(1H-1,2,4-triazol-1-yl)-4-(3,4,5-trimethoxybenzoyl)phenyl)thiazol-2-yl)-2-amino-3-methylbutanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CKD-516 inj (Experimental)
  Interventions: Drug: CKD-516 inj

INTERVENTIONS:
Drug: CKD-516 inj — 5.0 mg/2ml; 1.0, 2.0, 3.3, 5, 7, 9 ~ mg/m2; Day 1, Day 8 every 3 weeks
  Other Names: CKD-516

SUMMARY:
A phase I study is conducted to determine the maximum tolerated dose (MTD), dose limiting toxicity (DLT), safety and pharmacokinetics (PK) profile of a single agent CKD-516 injection on a weekly schedule in patients with advanced solid cancers failed to standard therapy. The usefulness of the this regimen is evaluated by response rate, progression free survival and vascular disruption effect by Dynamic Contrast-Enhanced MRI (DCE-MRI).

DETAILED DESCRIPTION:
OBJECTIVES:

* I. Determine the maximum tolerated dose of CKD-516 administered at single doses every 21 days in patients with advanced solid tumors.
* II. Determine both the toxicity and dose limiting toxicity of this regimen in these patients.
* III. Determine the plasma and urine pharmacokinetics of CKD-516.
* IV. Gather preliminary data regarding possible antitumor effects in those patients with measurable diseae. Assess the effects of CKD-516 on tumor blood flow using DCE-MRI scanning techniques, and establish the dose at which these effects occur.

OUTLINE: This is an open label, dose escalation study. Patients receive CKD-516 IV over 30 minutes on day 1, 8 every 3 weeks in the absence of unacceptable toxicity or disease progression. Cohorts of 3~6 patients receive escalating doses of CKD-516 until the maximum tolerated dose(MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 20~75 years
* Histologically or cytologically confirmed solid tumors that have failed to standard therapy or for which no life prolonging treatment exists
* ECOG PS 0-2
* Life expectancy 12 weeks
* Hematopoietic: ANC ≥ 1,500/mm3, Platelet ≥ 100,000/mm3, Hemoglobin ≥ 9.0g/dL, Prothrombin time, Activated partial thromboplastin time: normal range
* Hepatic: total bilirubin ≤ 1.5×ULN(except Gilbert's syndrome patients), AST, ALT ≤ 3.0×ULN(AST, ALT ≤ 5.0×ULN in case of liver metastases)
* Renal: serum creatinine ≤ 1.5×ULN or Creatinine clearance ≥ 60 mL/min
* Signed a written informed consent

Exclusion Criteria:

* Brain or Leptomeningeal metastases
* History of Ischemic heart disease(e.g., myocardial infarction, unstable angina pectoris) or Clinically significant heart disease such as NYHA Class III and IV Congestive atrial arrhythmias, within 6 months prior to first dose of study drug
* Stable angina pectoris shown symptoms within 6 months prior to first dose of study durg, or Clinically significant abnormality on EKG or echocardiogram(e.g., LVEF < 50% or clinically significant heart wall abnormality or heart muscle damage)
* Cerebrovascular disease such as stroke
* Grade 2 or greater motor or sensory peripheral neuropathy
* Clinically significant eye diseases(e.g., Glaucoma or Proliferative diabetic retinopathy, Atrophic macular degeneration), or other clinically significant abnormality on screening visit
* Uncontrolled hypertension(greater than 150 mmHg systolic anc 100 mmHg diastolic regardless of medication)
* acute infection or blooding tendencies that would preclude study compliance
* Serious vascular disease such as Aortic aneurysm
* Other psychiatric disorders or other conditions that would preclude study compliance
* Receiving anticoagulation with warfarin, heparin, etc.
* Receiving antitumor therapy(surgery, immunotherapy or chemotherapy) within 4 weeks prior to first dose of study drug(6 weeks for nitrosoureas and mitomycin C, 2 weeks for radiation therapy)
* Other concurrent antitumor therapy
* History of Serious hypersensitivity or allergy
* Pregnant or nursing, active serum pregnancy test. Fertile patients must use effective contraception
* Participation in a clinical trial within 4 weeks of first dose of study drug

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
MTD, Maximum Tolerated Dose | 1st cycle
PK parameters of CKD-516 and its metabolite, S516, when CKD-516 administered on Days 1 and 8 of a 21-day cycle | 1st cycle
Dose-limiting Toxicity | 1st cycle

SECONDARY OUTCOMES:
ORR%, Objective response rate | every 2 cycle
PFS, Progression Free Survival | 30 days before or after last patient out
Vascular disruption effect(with DCE-MRI) | 24hr after 1st cycle day 1 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, MD., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KW, Lee JM, Jeon YS, Kang SE, Baek JH, Han JK, Choi BI, Bang YJ, Kiefer B, Block KT, Ji H, Bauer S, Kim C. Free-breathing dynamic contrast-enhanced MRI of the abdomen and chest using a radial gradient echo sequence with K-space weighted image contrast (KWIC). Eur Radiol. 2013 May;23(5):1352-60. doi: 10.1007/s00330-012-2699-4. Epub 2012 Nov 28. PMID 23187728